CLINICAL TRIAL: NCT01245933
Title: Impact of Systemic Manifestations/Comorbidities on Clinical State, Prognosis and Utilisation of Health Care Resources in Patients With COPD
Brief Title: Impact of Systemic Manifestations/Comorbidities on Clinical State, Prognosis, Utilisation of Health Care Resources in Patients With COPD
Acronym: COSYCONET
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Collaborators: Hannover Medical School (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Claus Vogelmeier, Prof. Dr., Philipps University Marburg
Other Study IDs: 01GI0881
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; register; comorbidities; systemic inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood urine sputum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the prevalence and severity of extrapulmonary disorders and to quantify the impact of extrapulmonary organ manifestations on morbidity and mortality of COPD patients.

Furthermore the investigators evaluate the relationship between systemic inflammation and organ involvement.

DETAILED DESCRIPTION:
Chronic diseases and comorbidities have an increasing impact on individual life and health care use, as exemplified in chronic obstructive pulmonary disease (COPD). Currently, independent, comprehensive databases allowing for an integrated view are lacking. The study will for the first time establish a large, comprehensive longitudinal database covering a broad panel of comorbidities an markers of systemic alterations. These data will be of unique value in revealing specific phenotypes of COPD via patterns and risk profiles of comorbidities, enabling a more precise diagnosis and targeting of therapy, and an efficient allocation of resources.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 years and older
* diagnosis of COPD (GOLD-Criteria) or chronic bronchitis
* informed consent
* available for repeated study visits pver 18 months

Exclusion Criteria:

* having undergone big lung surgery (e.g. lung reduction, lung transplant)
* Moderate or severe exacerbation within the last 4 weeks
* having a lung tumor
* Unable to walk or to understand the intention of the project

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since the original recruitment strategy was not as successful as expected,the mode of recruitment was extended to other physicians, patients' groups and organisations and advertising to local media. The recruitment is supported by professional measures of communication organized by the coordinating centre Marburg.
Sampling Method: Non-Probability Sample
Enrollment: 2741 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BODE-Score at 18 months | at initial visite, after 18, 36, 54, 72, 90 and 108 months
  The BODE-Score comprises BMI, airway obstruction, dyspnea and exercise capacity and is a good predictor for death in COPD patients. Progression is defined as a change in BODE-score by >=1 point over the observation period.

SECONDARY OUTCOMES:
COPD related mortality | after 18 months
  The rate of mortality was elevated after 6, 18, 36, 54, 72, 90 and 108 months
COPD related hospitalization | after 18, 36, 54, 72, 90 and 108 months
  The rate of hospitalizations was elevated in every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Vogelmeier, Prof., Study Chair — Philipps University Marburg
Locations (22):
- Germany (22):
  - Ev. Lungenklinik (ELK), Krankenhausbetriebs gGmbH, Pneumologische Klinik, Berlin
  - Forschungszentrum Borstel, Medizinische Klinik, Borstel
  - Klinik Donaustauf, Zentrum für Pneumologie, Donaustauf
  - Ruhrlandklinik Essen, Westdeutsches Lungenzentrum, Essen
  - EvA-Study Center, Helholtz Zentrum München, Gauting
  - Justus-Liebig-Universität, Medizinische Klinik II, Giessen
  - Universitätsklinikum Greifswald der Ernst-Moritz-Arndt Universität, Zentrum für Innere Medizin, Greifswald
  - Krankenhaus Großhansdorf, Pneumologisches Forschungsinstitut, Großhansdorf
  - HIT-Hamburger Institut für Therapieforschung GmbH, Hamburg
  - Medical School Hannover, Dep. of Pneumology, Hanover
  - Thoraxklinik Heidelberg, Heidelberg
  - University of Saarland, Homburg
  - Fachklinik für Lungenerkrankungen Philippsstiftung ev., Immenhausen
  - Universitiy of Kiel, Kiel
  - Universitätsklinikum Leipzig, Department Innere Medizin, Leipzig
  - Philipps-University Marburg, Medical Center, Dep. of Pneumology, Marburg
  - Ludwig-Maximilians-University, Medizinische Klinik Innenstadt, Munich
  - Klinikum Nürnberg, Medizinische Klinik 3, Schwerpunkt Pneumologie, Allergologie und Schlafmedizin, Nuremberg
  - Universitätsklinikum Rostock, Zentrum für Innere Medizin, Abt. f. Pneumologie, Rostock
  - Klinikum Berchtesgardener Land, Schön Kliniken, Fachzentrum für Pneumologie, Allergologie und Schlafmedizin, Schönau am Königssee
  - Krankenhaus Bethanien gGmbH, Solingen
  - Missionsärztliche Klinik GmbH, Innere Medizin, Würzburg

REFERENCES:
- [Background] Jorres RA, Welte T, Bals R, Koch A, Schnoor M, Vogelmeier C. [Systemic manifestations and comorbidities in patients with chronic obstructive pulmonary disease (COPD) and their effect on clinical state and course of the disease--an overview of the cohort study COSYCONET]. Dtsch Med Wochenschr. 2010 Mar;135(10):446-9. doi: 10.1055/s-0030-1249185. Epub 2010 Mar 2. German. PMID 20198540
- [Result] Wacker ME, Jorres RA, Schulz H, Heinrich J, Karrasch S, Karch A, Koch A, Peters A, Leidl R, Vogelmeier C, Holle R; COSYCONET-Consortium. Direct and indirect costs of COPD and its comorbidities: Results from the German COSYCONET study. Respir Med. 2016 Feb;111:39-46. doi: 10.1016/j.rmed.2015.12.001. Epub 2015 Dec 10. PMID 26725462
- [Result] Karch A, Vogelmeier C, Welte T, Bals R, Kauczor HU, Biederer J, Heinrich J, Schulz H, Glaser S, Holle R, Watz H, Korn S, Adaskina N, Biertz F, Vogel C, Vestbo J, Wouters EF, Rabe KF, Sohler S, Koch A, Jorres RA; COSYCONET Study Group. The German COPD cohort COSYCONET: Aims, methods and descriptive analysis of the study population at baseline. Respir Med. 2016 May;114:27-37. doi: 10.1016/j.rmed.2016.03.008. Epub 2016 Mar 11. PMID 27109808
- [Result] Wacker ME, Jorres RA, Karch A, Wilke S, Heinrich J, Karrasch S, Koch A, Schulz H, Watz H, Leidl R, Vogelmeier C, Holle R; COSYCONET-Consortium. Assessing health-related quality of life in COPD: comparing generic and disease-specific instruments with focus on comorbidities. BMC Pulm Med. 2016 May 10;16(1):70. doi: 10.1186/s12890-016-0238-9. PMID 27160582
- [Result] Wacker ME, Jorres RA, Karch A, Koch A, Heinrich J, Karrasch S, Schulz H, Peters A, Glaser S, Ewert R, Baumeister SE, Vogelmeier C, Leidl R, Holle R; COSYCONET study group. Relative impact of COPD and comorbidities on generic health-related quality of life: a pooled analysis of the COSYCONET patient cohort and control subjects from the KORA and SHIP studies. Respir Res. 2016 Jul 12;17(1):81. doi: 10.1186/s12931-016-0401-0. PMID 27405652
- [Result] Lucke T, Herrera R, Wacker M, Holle R, Biertz F, Nowak D, Huber RM, Sohler S, Vogelmeier C, Ficker JH, Muckter H, Jorres RA; COSYCONET-Consortium. Systematic Analysis of Self-Reported Comorbidities in Large Cohort Studies - A Novel Stepwise Approach by Evaluation of Medication. PLoS One. 2016 Oct 28;11(10):e0163408. doi: 10.1371/journal.pone.0163408. eCollection 2016. PMID 27792735
- [Result] Alter P, Watz H, Kahnert K, Pfeifer M, Randerath WJ, Andreas S, Waschki B, Kleibrink BE, Welte T, Bals R, Schulz H, Biertz F, Young D, Vogelmeier CF, Jorres RA. Airway obstruction and lung hyperinflation in COPD are linked to an impaired left ventricular diastolic filling. Respir Med. 2018 Apr;137:14-22. doi: 10.1016/j.rmed.2018.02.011. Epub 2018 Feb 19. PMID 29605197
- [Result] Kahnert K, Lucke T, Huber RM, Behr J, Biertz F, Vogt A, Watz H, Alter P, Fahndrich S, Bals R, Holle R, Karrasch S, Sohler S, Wacker M, Ficker JH, Parhofer KG, Vogelmeier C, Jorres RA; COSYCONET consortium. Relationship of hyperlipidemia to comorbidities and lung function in COPD: Results of the COSYCONET cohort. PLoS One. 2017 May 15;12(5):e0177501. doi: 10.1371/journal.pone.0177501. eCollection 2017. PMID 28505167
- [Result] Fahndrich S, Biertz F, Karch A, Kleibrink B, Koch A, Teschler H, Welte T, Kauczor HU, Janciauskiene S, Jorres RA, Greulich T, Vogelmeier CF, Bals R; COSYCONET investigators. Cardiovascular risk in patients with alpha-1-antitrypsin deficiency. Respir Res. 2017 Sep 15;18(1):171. doi: 10.1186/s12931-017-0655-1. PMID 28915894
- [Result] Kahnert K, Alter P, Young D, Lucke T, Heinrich J, Huber RM, Behr J, Wacker M, Biertz F, Watz H, Bals R, Welte T, Wirtz H, Herth F, Vestbo J, Wouters EF, Vogelmeier CF, Jorres RA. The revised GOLD 2017 COPD categorization in relation to comorbidities. Respir Med. 2018 Jan;134:79-85. doi: 10.1016/j.rmed.2017.12.003. Epub 2017 Dec 5. PMID 29413512
- [Result] Kahnert K, Lucke T, Biertz F, Lechner A, Watz H, Alter P, Bals R, Behr J, Holle R, Huber RM, Karrasch S, Stubbe B, Wacker M, Sohler S, Wouters EF, Vogelmeier C, Jorres RA; COSYCONET study group. Transfer factor for carbon monoxide in patients with COPD and diabetes: results from the German COSYCONET cohort. Respir Res. 2017 Jan 13;18(1):14. doi: 10.1186/s12931-016-0499-0. PMID 28086884
- [Result] Houben-Wilke S, Jorres RA, Bals R, Franssen FM, Glaser S, Holle R, Karch A, Koch A, Magnussen H, Obst A, Schulz H, Spruit MA, Wacker ME, Welte T, Wouters EF, Vogelmeier C, Watz H. Peripheral Artery Disease and Its Clinical Relevance in Patients with Chronic Obstructive Pulmonary Disease in the COPD and Systemic Consequences-Comorbidities Network Study. Am J Respir Crit Care Med. 2017 Jan 15;195(2):189-197. doi: 10.1164/rccm.201602-0354OC. PMID 27532739
- [Result] Karl FM, Holle R, Bals R, Greulich T, Jorres RA, Karch A, Koch A, Karrasch S, Leidl R, Schulz H, Vogelmeier C, Wacker ME; COSYCONET Study Group. Costs and health-related quality of life in Alpha-1-Antitrypsin Deficient COPD patients. Respir Res. 2017 Apr 17;18(1):60. doi: 10.1186/s12931-017-0543-8. PMID 28416015
- [Result] Smid DE, Franssen FME, Gonik M, Miravitlles M, Casanova C, Cosio BG, de Lucas-Ramos P, Marin JM, Martinez C, Mir I, Soriano JB, de Torres JP, Agusti A, Atalay NB, Billington J, Boutou AK, Brighenti-Zogg S, Chaplin E, Coster S, Dodd JW, Durr S, Fernandez-Villar A, Groenen MTJ, Guimaraes M, Hejduk K, Higgins V, Hopkinson NS, Horita N, Houben-Wilke S, Janssen DJA, Jehn M, Joerres R, Karch A, Kelly JL, Kim YI, Kimura H, Koblizek V, Kocks JH, Kon SSC, Kwon N, Ladeira I, Lee SD, Leuppi JD, Locantore N, Lopez-Campos JL, D-C Man W, Maricic L, Mendoza L, Miedinger D, Mihaltan F, Minami S, van der Molen T, Murrells TJ, Nakken N, Nishijima Y, Norman IJ, Novotna B, O'Donnell DE, Ogata Y, Pereira ED, Piercy J, Price D, Pothirat C, Raghavan N, Ringbaek T, Sajkov D, Sigari N, Singh S, Small M, da Silva GF, Tanner RJ, Tsiligianni IG, Tulek B, Tzanakis N, Vanfleteren LEGW, Watz H, Webb KA, Wouters EFM, Xie GG, Yoshikawa M, Spruit MA. Redefining Cut-Points for High Symptom Burden of the Global Initiative for Chronic Obstructive Lung Disease Classification in 18,577 Patients With Chronic Obstructive Pulmonary Disease. J Am Med Dir Assoc. 2017 Dec 1;18(12):1097.e11-1097.e24. doi: 10.1016/j.jamda.2017.09.003. PMID 29169740
- [Result] Wacker ME, Kitzing K, Jorres RA, Leidl R, Schulz H, Karrasch S, Karch A, Koch A, Vogelmeier CF, Holle R. The contribution of symptoms and comorbidities to the economic impact of COPD: an analysis of the German COSYCONET cohort. Int J Chron Obstruct Pulmon Dis. 2017 Dec 4;12:3437-3448. doi: 10.2147/COPD.S141852. eCollection 2017. PMID 29270005
- [Result] Alter P, Jorres RA, Watz H, Welte T, Glaser S, Schulz H, Bals R, Karch A, Wouters EFM, Vestbo J, Young D, Vogelmeier CF. Left ventricular volume and wall stress are linked to lung function impairment in COPD. Int J Cardiol. 2018 Jun 15;261:172-178. doi: 10.1016/j.ijcard.2018.02.074. PMID 29657040
- [Result] Alter P, Rabe KF, Schulz H, Vogelmeier CF, Jorres RA. Influence of body mass on predicted values of static hyperinflation in COPD. Int J Chron Obstruct Pulmon Dis. 2018 Aug 23;13:2551-2555. doi: 10.2147/COPD.S164096. eCollection 2018. PMID 30197511
- [Result] Alter P, Jorres RA. Concomitance of cardiovascular and pulmonary disorders: mutual bystanders or causal interactions? Kardiol Pol. 2018;76(7):1027-1028. doi: 10.5603/KP.2018.0132. No abstract available. PMID 29984808
- [Result] Graf J, Lucke T, Herrera R, Watz H, Holle R, Vogelmeier C, Ficker JH, Jorres RA. Compatibility of medication with PRISCUS criteria and identification of drug interactions in a large cohort of patients with COPD. Pulm Pharmacol Ther. 2018 Apr;49:123-129. doi: 10.1016/j.pupt.2018.01.011. Epub 2018 Feb 5. PMID 29421666
- [Result] Graf J, Jorres RA, Lucke T, Nowak D, Vogelmeier CF, Ficker JH. Medical Treatment of COPD. Dtsch Arztebl Int. 2018 Sep 14;155(37):599-605. doi: 10.3238/arztebl.2018.0599. PMID 30282573
- [Result] Greulich T, Mager S, Lucke T, Koczulla AR, Bals R, Fahndrich S, Jorres RA, Alter P, Kirsten A, Vogelmeier CF, Watz H. Longitudinal stability of blood eosinophil count strata in the COPD COSYCONET cohort. Int J Chron Obstruct Pulmon Dis. 2018 Sep 28;13:2999-3002. doi: 10.2147/COPD.S165909. eCollection 2018. No abstract available. PMID 30319247
- [Result] Kahnert K, Alter P, Welte T, Huber RM, Behr J, Biertz F, Watz H, Bals R, Vogelmeier CF, Jorres RA. Uric acid, lung function, physical capacity and exacerbation frequency in patients with COPD: a multi-dimensional approach. Respir Res. 2018 Jun 4;19(1):110. doi: 10.1186/s12931-018-0815-y. PMID 29866121
- [Result] Kahnert K, Jobst B, Biertz F, Biederer J, Watz H, Huber RM, Behr J, Grenier PA, Alter P, Vogelmeier CF, Kauczor HU, Jorres RA. Relationship of spirometric, body plethysmographic, and diffusing capacity parameters to emphysema scores derived from CT scans. Chron Respir Dis. 2019 Jan-Dec;16:1479972318775423. doi: 10.1177/1479972318775423. Epub 2018 May 9. PMID 29742906
- [Result] Kaireit TF, Voskrebenzev A, Gutberlet M, Freise J, Jobst B, Kauczor HU, Welte T, Wacker F, Vogel-Claussen J. Comparison of quantitative regional perfusion-weighted phase resolved functional lung (PREFUL) MRI with dynamic gadolinium-enhanced regional pulmonary perfusion MRI in COPD patients. J Magn Reson Imaging. 2019 Apr;49(4):1122-1132. doi: 10.1002/jmri.26342. Epub 2018 Oct 22. PMID 30350440
- [Result] Keller A, Fehlmann T, Ludwig N, Kahraman M, Laufer T, Backes C, Vogelmeier C, Diener C, Biertz F, Herr C, Jorres RA, Lenhof HP, Meese E, Bals R; COSYCONET Study Group. Genome-wide MicroRNA Expression Profiles in COPD: Early Predictors for Cancer Development. Genomics Proteomics Bioinformatics. 2018 Jun;16(3):162-171. doi: 10.1016/j.gpb.2018.06.001. Epub 2018 Jul 5. PMID 29981854
- [Result] Triphan SMF, Biederer J, Burmester K, Fellhauer I, Vogelmeier CF, Jorres RA, Kauczor HU, Heussel CP, Wielputz MO, Jobst BJ. Design and application of an MR reference phantom for multicentre lung imaging trials. PLoS One. 2018 Jul 5;13(7):e0199148. doi: 10.1371/journal.pone.0199148. eCollection 2018. PMID 29975714
- [Result] Alter P, Watz H, Kahnert K, Rabe KF, Biertz F, Fischer R, Jung P, Graf J, Bals R, Vogelmeier CF, Jorres RA. Effects of airway obstruction and hyperinflation on electrocardiographic axes in COPD. Respir Res. 2019 Mar 27;20(1):61. doi: 10.1186/s12931-019-1025-y. PMID 30917825
- [Result] Byng D, Lutter JI, Wacker ME, Jorres RA, Liu X, Karrasch S, Schulz H, Vogelmeier C, Holle R. Determinants of healthcare utilization and costs in COPD patients: first longitudinal results from the German COPD cohort COSYCONET. Int J Chron Obstruct Pulmon Dis. 2019 Jul 5;14:1423-1439. doi: 10.2147/COPD.S201899. eCollection 2019. PMID 31308648
- [Result] Trudzinski FC, Kahnert K, Vogelmeier CF, Alter P, Seiler F, Fahndrich S, Watz H, Welte T, Speer T, Zewinger S, Biertz F, Kauczor HU, Jorres RA, Bals R; COSYCONET consortium. Combined effects of lung function, blood gases and kidney function on the exacerbation risk in stable COPD: Results from the COSYCONET cohort. Respir Med. 2019 Jul-Aug;154:18-26. doi: 10.1016/j.rmed.2019.06.007. Epub 2019 Jun 11. PMID 31203096
- [Result] Trudzinski FC, Alqudrah M, Omlor A, Zewinger S, Fliser D, Speer T, Seiler F, Biertz F, Koch A, Vogelmeier C, Welte T, Watz H, Waschki B, Fahndrich S, Jorres R, Bals R; German COSYCONET consortium. Consequences of chronic kidney disease in chronic obstructive pulmonary disease. Respir Res. 2019 Jul 12;20(1):151. doi: 10.1186/s12931-019-1107-x. PMID 31299972
- [Result] von Siemens SM, Jorres RA, Behr J, Alter P, Lutter J, Lucke T, Sohler S, Welte T, Watz H, Vogelmeier CF, Trudzinski F, Rief W, Herbig B, Kahnert K; COSYCONET study group. Effect of COPD severity and comorbidities on the result of the PHQ-9 tool for the diagnosis of depression: results from the COSYCONET cohort study. Respir Res. 2019 Feb 11;20(1):30. doi: 10.1186/s12931-019-0997-y. PMID 30744630
- [Result] Alter P, Mayerhofer BA, Kahnert K, Watz H, Waschki B, Andreas S, Biertz F, Bals R, Vogelmeier CF, Jorres RA. Prevalence of cardiac comorbidities, and their underdetection and contribution to exertional symptoms in COPD: results from the COSYCONET cohort. Int J Chron Obstruct Pulmon Dis. 2019 Sep 20;14:2163-2172. doi: 10.2147/COPD.S209343. eCollection 2019. PMID 31571852
- [Result] Keller A, Ludwig N, Fehlmann T, Kahraman M, Backes C, Kern F, Vogelmeier CF, Diener C, Fischer U, Biertz F, Herr C, Jorres RA, Lenhof HP, Bals R, Meese E. Low miR-150-5p and miR-320b Expression Predicts Reduced Survival of COPD Patients. Cells. 2019 Sep 27;8(10):1162. doi: 10.3390/cells8101162. PMID 31569706
- [Result] Konigsdorfer N, Jorres RA, Sohler S, Welte T, Behr J, Ficker JH, Bals R, Watz H, Lutter JI, Lucke T, Biertz F, Alter P, Vogelmeier CF, Kahnert K. Adherence To Respiratory And Nonrespiratory Medication In Patients With COPD: Results Of The German COSYCONET Cohort. Patient Prefer Adherence. 2019 Oct 10;13:1711-1721. doi: 10.2147/PPA.S223438. eCollection 2019. PMID 31631986
- [Result] von Siemens SM, Perneczky R, Vogelmeier CF, Behr J, Kauffmann-Guerrero D, Alter P, Trudzinski FC, Bals R, Grohe C, Sohler S, Waschki B, Lutter JI, Welte T, Jorres RA, Kahnert K; COSYCONET study group. The association of cognitive functioning as measured by the DemTect with functional and clinical characteristics of COPD: results from the COSYCONET cohort. Respir Res. 2019 Nov 14;20(1):257. doi: 10.1186/s12931-019-1217-5. PMID 31727165
- [Result] Kahnert K, Fohrenbach M, Lucke T, Alter P, Trudzinski FT, Bals R, Lutter JI, Timmermann H, Sohler S, Forderreuther S, Nowak D, Watz H, Waschki B, Behr J, Welte T, Vogelmeier CF, Jorres RA. The impact of COPD on polyneuropathy: results from the German COPD cohort COSYCONET. Respir Res. 2020 Jan 20;21(1):28. doi: 10.1186/s12931-020-1293-6. PMID 31959163
- [Result] Lutter JI, Jorres RA, Kahnert K, Schwarzkopf L, Studnicka M, Karrasch S, Schulz H, Vogelmeier CF, Holle R; COSYCONET Study Group. Health-related quality of life associates with change in FEV1 in COPD: results from the COSYCONET cohort. BMC Pulm Med. 2020 May 29;20(1):148. doi: 10.1186/s12890-020-1147-5. PMID 32471493
- [Result] Trudzinski FC, Jorres RA, Alter P, Kahnert K, Waschki B, Herr C, Kellerer C, Omlor A, Vogelmeier CF, Fahndrich S, Watz H, Welte T, Jany B, Sohler S, Biertz F, Herth F, Kauczor HU, Bals R; COSYCONET consortium. Associations of oxygenated hemoglobin with disease burden and prognosis in stable COPD: Results from COSYCONET. Sci Rep. 2020 Jun 29;10(1):10544. doi: 10.1038/s41598-020-67197-x. PMID 32601330
- [Result] Marietta von Siemens S, Alter P, Lutter JI, Kauczor HU, Jobst B, Bals R, Trudzinski FC, Sohler S, Behr J, Watz H, Waschki B, Bewig B, Jones PW, Welte T, Vogelmeier CF, Jorres RA, Kahnert K; COSYCONET study group; Names of participating study nurses. CAT score single item analysis in patients with COPD: Results from COSYCONET. Respir Med. 2019 Nov;159:105810. doi: 10.1016/j.rmed.2019.105810. Epub 2019 Nov 7. PMID 31739262
- [Result] Lutter JI, Lukas M, Schwarzkopf L, Jorres RA, Studnicka M, Kahnert K, Karrasch S, Bewig B, Vogelmeier CF, Holle R; COSYCONET Study Group. Utilization and determinants of use of non-pharmacological interventions in COPD: Results of the COSYCONET cohort. Respir Med. 2020 Sep;171:106087. doi: 10.1016/j.rmed.2020.106087. Epub 2020 Jul 12. PMID 32917358
- [Result] Waschki B, Alter P, Zeller T, Magnussen C, Neumann JT, Twerenbold R, Sinning C, Herr C, Kahnert K, Fahndrich S, Blankenberg S, Rabe KF, Welte T, Jorres RA, Vogelmeier CF, Bals R, Watz H; German COSYCONET Cohort. High-sensitivity troponin I and all-cause mortality in patients with stable COPD: an analysis of the COSYCONET study. Eur Respir J. 2020 Feb 27;55(2):1901314. doi: 10.1183/13993003.01314-2019. Print 2020 Feb. PMID 31831579
- [Result] Omlor AJ, Trudzinski FC, Alqudrah M, Seiler F, Biertz F, Vogelmeier CF, Welte T, Watz H, Waschki B, Brinker TJ, Andreas S, Fahndrich S, Alter P, Jorres RA, Bohm M, Bals R; German COSYCONET Cohort. Time-updated resting heart rate predicts mortality in patients with COPD. Clin Res Cardiol. 2020 Jun;109(6):776-786. doi: 10.1007/s00392-019-01572-1. Epub 2019 Nov 16. PMID 31734762
- [Result] Lommatzsch M, Speer T, Herr C, Jorres RA, Watz H, Muller A, Welte T, Vogelmeier CF, Bals R; COSYCONET study group. IgE is associated with exacerbations and lung function decline in COPD. Respir Res. 2022 Jan 4;23(1):1. doi: 10.1186/s12931-021-01847-0. PMID 34983515
- [Result] Kellerer C, Jorres RA, Schneider A, Alter P, Kauczor HU, Jobst B, Biederer J, Bals R, Watz H, Behr J, Kauffmann-Guerrero D, Lutter J, Hapfelmeier A, Magnussen H, Trudzinski FC, Welte T, Vogelmeier CF, Kahnert K. Prediction of lung emphysema in COPD by spirometry and clinical symptoms: results from COSYCONET. Respir Res. 2021 Sep 9;22(1):242. doi: 10.1186/s12931-021-01837-2. PMID 34503520
- [Result] Trudzinski FC, Jorres RA, Alter P, Walter J, Watz H, Koch A, John M, Lommatzsch M, Vogelmeier CF, Kauczor HU, Welte T, Behr J, Tufman A, Bals R, Herth FJF, Kahnert K; COSYCONET Study Group. Sex-specific associations of comorbidome and pulmorbidome with mortality in chronic obstructive pulmonary disease: results from COSYCONET. Sci Rep. 2022 May 24;12(1):8790. doi: 10.1038/s41598-022-12828-8. PMID 35610473
- [Derived] Alter P, Watz H, Machado FVC, Speicher T, Trudzinski FC, Kahnert K, Bals R, Wouters EFM, Franssen FME, Vogelmeier CF, Karrasch S, Jorres RA. Association of Obesity with Symptoms and Quality of Life in COPD: Results from COSYCONET. Int J Chron Obstruct Pulmon Dis. 2025 Dec 25;20:4129-4141. doi: 10.2147/COPD.S542628. eCollection 2025. PMID 41476636
- [Derived] Eichenlaub M, Frye BC, Lehrmann H, Biertz F, Jadidi AS, Kaier K, Melzer T, Alter P, Watz H, Waschki B, Weckler BC, Trudzinski FC, Michels-Zetsche JD, Trinkmann F, Herth FJ, Kauczor HU, Kahnert K, Jorres R, Bals R, Westermann D, Arentz T, Vogelmeier CF, Stolz D, Fahndrich S; German COSYCONET cohort. ECG-based identification of COPD patients at risk for atrial fibrillation and its impact on adverse clinical outcomes-a subgroup analysis of the prospective multicenter COSYCONET cohort. Respir Res. 2025 Sep 17;26(1):272. doi: 10.1186/s12931-025-03342-2. PMID 40963108
- [Derived] Alter P, Kahnert K, Trudzinski FC, Bals R, Watz H, Speicher T, Sohler S, Rabe KF, Wouters EFM, Vogelmeier CF, Jorres RA. Unravelling the Information Contained in the Single Items of the COPD Assessment Test for Different Outcomes and Smoking Status in Patients with COPD: Results from COSYCONET. Int J Chron Obstruct Pulmon Dis. 2024 Dec 5;19:2629-2638. doi: 10.2147/COPD.S475112. eCollection 2024. PMID 39655060
- [Derived] Trudzinski FC, Jorres RA, Alter P, Watz H, Vogelmeier CF, Kauczor HU, Thangamani S, Debic M, Welte T, Behr J, Kahnert K, Bals R, Herr C, Heussel CP, Biederer J, von Stackelberg O, Fahndrich S, Wouters EFM, Waschki B, Rabe KF, Herth FJF, Palm V; COSYCONET study group. Midregional Proatrial Natriuretic Peptide (MRproANP) is associated with vertebral fractures and low bone density in patients with chronic obstructive pulmonary disease (COPD). Respir Res. 2024 Jul 13;25(1):274. doi: 10.1186/s12931-024-02902-2. PMID 39003487
- [Derived] Abdo M, Watz H, Alter P, Kahnert K, Trudzinski F, Groth EE, Claussen M, Kirsten AM, Welte T, Jorres RA, Vogelmeier CF, Bals R, Rabe KF, Waschki B. Characterization and Mortality Risk of Impaired Left Ventricular Filling in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2025 Mar;211(3):477-485. doi: 10.1164/rccm.202310-1848OC. PMID 38984876
- [Derived] Stoleriu MG, Pienn M, Joerres RA, Alter P, Fero T, Urschler M, Kovacs G, Olschewski H, Kauczor HU, Wielputz M, Jobst B, Welte T, Behr J, Trudzinski FC, Bals R, Watz H, Vogelmeier CF, Biederer J, Kahnert K; COSYCONET Study Group. Expiratory Venous Volume and Arterial Tortuosity are Associated with Disease Severity and Mortality Risk in Patients with COPD: Results from COSYCONET. Int J Chron Obstruct Pulmon Dis. 2024 Jul 1;19:1515-1529. doi: 10.2147/COPD.S458905. eCollection 2024. PMID 38974817
- [Derived] Frantzi N, Nguyen XP, Herr C, Alter P, Sohler S, Soriano D, Watz H, Waschki B, Trinkmann F, Eichenlaub M, Trudzinski FC, Michels-Zetsche JD, Omlor A, Seiler F, Moneke I, Biertz F, Rohde G, Stolz D, Welte T, Kauczor HU, Kahnert K, Jorres RA, Vogelmeier CF, Bals R, Fahndrich S; German COSYCONET Cohort. Statins did not reduce the frequency of exacerbations in individuals with COPD and cardiovascular comorbidities in the COSYCONET cohort. Respir Res. 2024 May 15;25(1):207. doi: 10.1186/s12931-024-02822-1. PMID 38750572
- [Derived] Gerlich J, Ohlander J, Kromhout H, Vermeulen R, Sohler S, Radon K, Nowak D, Karrasch S, Adaskina N, Vogelmeier C, Ochmann U, Jorres RA. Cumulative occupational exposure to gases and fumes is associated with impairment in lung function and disease-related quality of life in a German COPD patient cohort. Occup Environ Med. 2023 Dec 30;81(1):26-33. doi: 10.1136/oemed-2023-108908. Online ahead of print. PMID 38160050
- [Derived] Alter P, Kahnert K, Trudzinski FC, Bals R, Watz H, Speicher T, Sohler S, Welte T, Rabe KF, Wouters EFM, Vogelmeier CF, Jorres RA. Clinical factors linked to the type of respiratory medication in COPD: results from the COSYCONET cohort. Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231208584. doi: 10.1177/17534666231208584. PMID 37936408
- [Derived] Kahnert K, Jorres RA, Kauczor HU, Alter P, Trudzinski FC, Herth F, Jobst B, Weinheimer O, Nauck S, Mertsch P, Kauffmann-Guerrero D, Behr J, Bals R, Watz H, Rabe KF, Welte T, Vogelmeier CF, Biederer J. Standardized airway wall thickness Pi10 from routine CT scans of COPD patients as imaging biomarker for disease severity, lung function decline, and mortality. Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666221148663. doi: 10.1177/17534666221148663. PMID 36718763
- [Derived] Alter P, Lucke T, Watz H, Andreas S, Kahnert K, Trudzinski FC, Speicher T, Sohler S, Bals R, Waschki B, Welte T, Rabe KF, Vestbo J, Wouters EFM, Vogelmeier CF, Jorres RA. Cardiovascular predictors of mortality and exacerbations in patients with COPD. Sci Rep. 2022 Dec 19;12(1):21882. doi: 10.1038/s41598-022-25938-0. PMID 36536050
- [Derived] Kahnert K, Jorres RA, Lucke T, Trudzinski FC, Mertsch P, Bickert C, Ficker JH, Behr J, Bals R, Watz H, Welte T, Vogelmeier CF, Alter P; COSYCONET Study Group. Lower Prevalence of Osteoporosis in Patients with COPD Taking Anti-Inflammatory Compounds for the Treatment of Diabetes: Results from COSYCONET. Int J Chron Obstruct Pulmon Dis. 2021 Nov 24;16:3189-3199. doi: 10.2147/COPD.S335029. eCollection 2021. PMID 34853511
- [Derived] Trudzinski FC, Kellerer C, Jorres RA, Alter P, Lutter JI, Trinkmann F, Herth FJF, Frankenberger M, Watz H, Vogelmeier CF, Kauczor HU, Welte T, Behr J, Bals R, Kahnert K. Gender-specific differences in COPD symptoms and their impact for the diagnosis of cardiac comorbidities. Clin Res Cardiol. 2023 Feb;112(2):177-186. doi: 10.1007/s00392-021-01915-x. Epub 2021 Jul 31. PMID 34331588
- [Derived] Kellerer C, Kahnert K, Trudzinski FC, Lutter J, Berschneider K, Speicher T, Watz H, Bals R, Welte T, Vogelmeier CF, Jorres RA, Alter P. COPD maintenance medication is linked to left atrial size: Results from the COSYCONET cohort. Respir Med. 2021 Aug-Sep;185:106461. doi: 10.1016/j.rmed.2021.106461. Epub 2021 May 29. PMID 34116329
- [Derived] Alter P, Orszag J, Kellerer C, Kahnert K, Speicher T, Watz H, Bals R, Welte T, Vogelmeier CF, Jorres RA. Prediction of air trapping or pulmonary hyperinflation by forced spirometry in COPD patients: results from COSYCONET. ERJ Open Res. 2020 Jul 27;6(3):00092-2020. doi: 10.1183/23120541.00092-2020. eCollection 2020 Jul. PMID 32743009
- See also: Description of the study, study results, links to relevant organisaton — http://www.asconet.net
- Available data/document: general information — http://www.asconet.net